CLINICAL TRIAL: NCT01381588
Title: The Prevalence of Osteoporotic Vertebral Compression Fractures (OVCF) in Korean Post Menopausal Women
Acronym: TOP
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114777
Record Dates: First submitted 2011-06-09; First posted 2011-06-27 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — X-Rays

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Post menopausal women: Post menopausal women between 50 to 80
  Interventions: Other: Fracture evaluation

INTERVENTIONS:
Other: Fracture evaluation — DEXA(Dual-energy X-ray absorptiometry), X-ray
  Other Names: X-ray

SUMMARY:
This is an observational study to investigate the prevalence of osteoporotic fractures in post menopausal patients. Post menopausal patients who visit OS(orthopedic surgery) including GHs(general hospitals) and clinics will be enrolled.

DETAILED DESCRIPTION:
This is an observational study to investigate the prevalence of osteoporotic fractures in post menopausal patients. Post menopausal patients who visit OS(orthopedic surgery) including GHs(general hospitals) and clinics will be enrolled. They will take the evaluation of spine X-ray and answer to a few questions. Their medical record will be reviewed and relevant clinical findings will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were diagnosed post menopausal state
* Subjects over 50 years old
* The Definition of Post Menopause Women : Women whose last menstruation was over 12months ago
* Subjects who visit orthopedic surgery
* Subjects who have informed consents

Exclusion Criteria:

* Subjects who are not confirmed as post menopause state
* Subjects who do not understand the contents of questionnaire
* Subjects over 80 years old
* Subjects experienced any high energy fracture (including trash and fall) within 3 months.
* Subjects experienced a fracture except vertebral fracture within 6 months
* Unable to evaluate L-spine BMD over 2 levels because of spinal fracture or instrumentation for L-spine 1-4.
* Unable to evaluate BMD at both femur because of hip fracture or instrumentation.

Ages: 50 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women
Sampling Method: Probability Sample
Enrollment: 1136 (Actual)
Dates: Start 2010-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
The prevalence of OVCFs confirmed by history and X-ray | 1 day

SECONDARY OUTCOMES:
The prevalence of asymptomatic (or missed) fractures | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Seoul, South Korea